CLINICAL TRIAL: NCT06910137
Title: An Early Access Program Guideline to Provide Access to Retifanlimab (INCMGA00012) Together With Carboplatin and Paclitaxel for Squamous Carcinoma of the Anal Canal (SCAC)
Status: Available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCMGA00012-EUMA-AC-301
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of the Anal Canal
Keywords: Squamous cell carcinoma; Anal Cancer; Retifanlimab; Expanded Access Program
MeSH Terms: conditions — Carcinoma, Squamous Cell; Anus Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: retifanlimab — Administered intravenous as defined in the protocol.
  Other Names: INCMGA00012

SUMMARY:
To provide retifanlimab, on a reactive basis, to adult patients with squamous carcinoma of the anal canal in combination with carboplatin and paclitaxel and who are considered ineligible for other therapeutic options including clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign a written ICF for the study.
* Are 18 years of age or older (or as applicable per local country requirements).
* Histologically or cytologically verified, inoperable locally recurrent or metastatic SCAC.
* Adequate ECOG performance status to be able to benefit from the treatment.
* If HIV-positive, a well controlled and stable disease and receiving antiretroviral therapy (ART/HAART) and have not experienced any HIV-related opportunistic infection for at least 4 weeks prior to study enrollment.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

  * Men must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through 120 days after the last dose of INCMGA00012 or placebo or through 180 days after the last dose of chemotherapeutic agents, whichever occurs later (or longer as appropriate based on country-specific requirements) and must refrain from donating sperm during this period. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Women of childbearing potential must have a negative serum pregnancy test at screening, agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty), and refrain from donating oocytes from screening through 120 days after the last dose of INCMGA00012 or placebo or through 180 days after the last dose of chemotherapeutic agents, whichever occurs later. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed. The definition of WOCBP is located in the protocol.
  * Women of nonchildbearing potential are eligible as defined in the protocol.

Exclusion Criteria:

* Has received prior PD-(L)1 directed therapy.
* Participants must have recovered from previous therapies for example including but not limited to RT and CRT.
* Participants with laboratory values at screening defined below:

Hematology:

* Platelets < 100 × 109/L.
* Hemoglobin < 9 g/dL.
* ANC < 1.5 x 109/L.

Hepatic:

* ALT ˃ 2.5 x ULN or ˃ 5 x ULN for participants with liver metastases.
* AST ˃ 2.5 x ULN or ˃ 5 x ULN for participants with liver metastases.
* Bilirubin ≥ 1.5 x ULN unless conjugated bilirubin ≤ ULN (conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN). If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin.

Renal:

• Calculated creatinine clearance < 50 mL/min calculated by Cockcroft-Gault equation (glomerular filtration rate can also be used in place of CrCl).

Coagulation:

* INR or PT > 1.5 × ULN, for participants not receiving anticoagulant therapy.
* aPTT > 1.5 × ULN for participants not receiving anticoagulant therapy.

  * Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg of prednisone or equivalent).
  * Evidence of interstitial lung disease or active noninfectious pneumonitis.
  * History of organ transplant, including allogeneic stem cell transplantation.
  * Known active CNS metastases and/or carcinomatous meningitis, per the protocol.
  * Known active HAV, HBV, or HCV infection, as defined by elevated transaminases with the following serology: positivity for HAV IgM antibody, anti-HCV, anti-HBc IgG or IgM, or HBsAg (in the absence of prior immunization).
  * Active infections requiring systemic therapy, or IV antibiotic use up to 7 days before Cycle 1 Day 1.
  * Known hypersensitivity to platinum, paclitaxel, another monoclonal antibody, or any of the excipients that cannot be controlled with standard measures (eg, antihistamines, corticosteroids).
  * Participants with impaired cardiac function or clinically significant cardiac disease as assessed by the treating physician.
  * Participant is pregnant or breastfeeding.
  * Has pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE v5.
  * Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: An Early Access Program Guideline to Provide Access to Retifanlimab (INCMGA00012) together with carboplatin and paclitaxel for Squamous Carcinoma of the Anal Canal (SCAC) — https://incyteclinicaltrials.com/studies/incmga00012-euma-ac-301